CLINICAL TRIAL: NCT01540565
Title: A Phase II Evaluation of the Poly (ADP-Ribose) Polymerase (PARP)-1 and -2 Inhibitor Veliparib (ABT-888) (NSC#737664) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients Who Carry a Germline BRCA1 or BRCA2 Mutation
Brief Title: Veliparib in Treating Patients With Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00684; NCI-2012-00684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S12-02446; GOG-0280; CDR0000726699; GOG-0280 (Other: NRG Oncology); GOG-0280 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-02-22; First posted 2012-02-29 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ovarian Epithelial Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (veliparib) (Experimental): Patients receive veliparib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase II trial studies how well veliparib works in treating patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer that has come back or does not respond to treatment. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who have objective tumor response (complete or partial).

II. To determine the frequency and severity of adverse events associated with treatment with veliparib (ABT-888) as assessed by the Active Version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival (PFS) and overall survival (OS).

II. To determine the proportion of patients who survive progression-free for at least 6 months.

TERTIARY OBJECTIVES:

I. To explore the association between single nucleotide polymorphisms (SNPs) in deoxyribonucleic acid (DNA) repair genes (e.g., breast cancer [BRCA]1, Fanconi) and clinical characteristics, response, and patient outcome (PFS and OS).

OUTLINE:

Patients receive veliparib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma AND carry a germline mutation in BRCA1 or BRCA2 (confirmation required via Myriad test report); histologic documentation of the original primary tumor is required via the pathology report
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors(RECIST)1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients who have received one prior cytotoxic regimen must have a Gynecological Oncology Group (GOG) performance status of 0, 1, or 2
* Patients who have received two or three prior cytotoxic regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted (non-cytotoxic) agents and immunologic agents, must be discontinued at least three weeks prior to registration; patients receiving nitrosoureas or mitomycin C must discontinue 6 weeks prior to registration
  * Any prior radiation therapy must be discontinued at least four weeks prior to registration
* Prior therapy

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents or extended therapy administered after surgical or non-surgical assessment
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease
  * Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy for management of recurrent or persistent disease; patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen
  * Patients with both platinum-sensitive and platinum-resistant disease are eligible; patients with platinum-refractory disease are NOT eligible
  * Definitions:

    * Platinum sensitive ovarian cancer is defined as patients who respond to platinum-based therapy (complete or partial) and then progress/recur more than 6 months after their last platinum dose (i.e., platinum-free interval is > 6 months)
    * Platinum resistant ovarian cancer is defined as patients who respond to platinum-based therapy (complete or partial) and then progress/recur within 6 months of their last platinum dose (i.e., platinum-free interval is =< 6 months)
    * Platinum refractory ovarian cancer is defined as patients who have progression of disease while receiving platinum-based chemotherapy or who fail to achieve at least a partial response to platinum-based chemotherapy (i.e., best response to platinum-based chemotherapy is stable disease)
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had previous treatment with veliparib (ABT-888) or any other poly (adenosine diphosphate [ADP]-ribose) polymerase 1 (PARP) inhibitor (including olaparib); note: Iniparib (BSI-201) cannot inhibit PARP1 at pharmacologically achievable concentrations, therefore prior iniparib therapy is allowed
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with seizures or history or seizures are ineligible
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, any CNS metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study are ineligible; patients with CNS metastases must be stable for > 3 months after treatment and off steroid treatment prior to study enrollment
* Inability or unwillingness to swallow pills
* Patients with clinical symptoms or signs of gastrointestinal obstruction and/or who require parenteral hydration or nutrition
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04-09 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — NRG Oncology
Locations (153):
- United States (153):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Gynecologic Oncology Associates-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to patient entry April 2012 and closed to accrual November 2012.
Period: Overall Study
Arm/Group | Treatment (Veliparib)
Started | 52
Completed | 50
Not Completed | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 2
  40-49 years | 15
  50-59 years | 14
  60-69 years | 15
  70-79 years | 2
  >=80 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 44
  More than one race | 0
  Unknown or Not Reported | 3
Cell Type [Count of Participants; unit: Participants]
  Serous | 41
  Other | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete and Partial Tumor Response
Description: Patients with complete and partial tumor response by RECIST V1.1 (per response evaluation criteria in Solid Tumors Criteria (RECIST V1.1) for target lesions and assessed by MRI (CT scan): Complete Response (CR), disappearance of all target lesions (confirmed at >= 4 weeks); Partial Response (PR) >= 30% decrease in the sum of the longest diameter of target lesions (confirmed at >= 4 weeks); Overall Response = CR + PR.
Time Frame: CT scan/MRI if used to follow lesion for measurable disease every other cycle for the first 6 months, then every 3 months until progression. Repeat at other times if clinically indicated.Responses require confirmation at >= 4 wks from first documentation.
Population: Eligible and evaluable
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
Proportion of patients | 0.26 [0.146 to 0.403]

2. Primary Outcome: Proportion of Patients With Adverse Events as Assessed by CTCAE v4.0
Description: Patients with grade 3 or greater Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Time Frame: After every cycle while on study therapy. Followed for late adverse events up to 30 days after completing therapy.
Population: Eligible and evaluable
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
Proportion of patients | 0.32 [0.195 to 0.467]

3. Secondary Outcome: Duration of PFS
Description: The time from randomization until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions (and >= 5 mm increase of target lesions), or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: CT scan/MRI if used to follow lesion for measurable disease every other cycle for the first 6 months, then every 3 months until progression. Patients who begin subsequent therapy without progression will be monitored for PFS for 5 years.
Population: Eligible and evaluable
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
months | 8.18 [5.45 to 9.63]

4. Secondary Outcome: Duration of OS
Description: Overall survival
Time Frame: Every cycle while patient is receiving protocol therapy. Patients will be monitored for survival after going off therapy for a 5 year period, every 3 months for the first 2 years, then every 6 months for the last 3 years.
Population: Eligible and evaluable
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
Months | NA [13.4 to NA] — The sample size was not sufficient for the calculation of the median. The first quartile of 13.4 months was calculated, but the data was not adequate for the computation of the median or the third quartile.

5. Secondary Outcome: The Proportion of Patients Who Survive Progression-free for at Least 6 Months
Description: This outcome captures whether or not the patient survived progression-free for at least 6 months, and is displayed as a proportion.
Time Frame: 6 months
Population: Eligible and evaluable
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 50
Proportion of patients | 0.54 [0.393 to 0.682]

6. Other Pre Specified Outcome: SNPs With DNA Repair Genes, Tumor Response, PFS, OS, and Patient Demographics (e.g. Age, Race, Tumor Grade)
Description: If the clinical trial goes to the second stage and there is sufficient variability in the SNPs, then patients can be categorized by the nature of their SNPs and assessed for prognostic value through survival analysis (e.g. log-rank tests and Cox proportional hazards modeling). If the variability in SNPs is relatively low, assessment of prognostic value can be conducted with odds ratios of patients responding or surviving progression-free for at least 6 months. These techniques will use exact methods such as Fisher's exact test.
Time Frame: Baseline
Population: Data not collected
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: BRCA Mutation in Primary Tumor Tissue
Description: BRCA mutational status will be tabulated against the germline mutation to see what proportion of patients have a mutation reversal within the tumor and whether such reversals can explain resistance to the regimen under study.
Time Frame: Baseline
Population: Data not collected
Arm/Group | Treatment (Veliparib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from study enrollment until 30 days after the last treatment, up to 5 years from enrollment.
Arm/Group | Treatment (Veliparib)
All-Cause Mortality (participants affected / at risk) | 21/50
Serious Adverse Events (participants affected / at risk) | 10/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Veliparib) (N=50)
Small Intestinal Obstruction (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Veliparib) (N=50)
Anemia (Blood and lymphatic system disorders) | 29
Palpitations (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 1
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 4
Hearing Impaired (Ear and labyrinth disorders) | 1
Watering Eyes (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 4
Colonic Perforation (Gastrointestinal disorders) | 1
Colonic Fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 33
Bloating (Gastrointestinal disorders) | 8
Stomach Pain (Gastrointestinal disorders) | 4
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 15
Periodontal Disease (Gastrointestinal disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 45
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Hemorrhoids (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Malaise (General disorders) | 4
Flu Like Symptoms (General disorders) | 6
Edema Trunk (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 4
Edema Limbs (General disorders) | 2
Fatigue (General disorders) | 35
Fever (General disorders) | 2
Chills (General disorders) | 2
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Enterocolitis Infectious (Infections and infestations) | 1
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 2
Weight Gain (Investigations) | 4
Platelet Count Decreased (Investigations) | 10
Lymphocyte Count Decreased (Investigations) | 8
Creatinine Increased (Investigations) | 3
Neutrophil Count Decreased (Investigations) | 18
Blood Bilirubin Increased (Investigations) | 3
White Blood Cell Decreased (Investigations) | 25
Aspartate Aminotransferase Increased (Investigations) | 8
Alkaline Phosphatase Increased (Investigations) | 9
Alanine Aminotransferase Increased (Investigations) | 9
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 1
Glucose Intolerance (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Tremor (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 14
Paresthesia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 3
Movements Involuntary (Nervous system disorders) | 2
Headache (Nervous system disorders) | 14
Dysgeusia (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 13
Depressed Level Of Consciousness (Nervous system disorders) | 1
Concentration Impairment (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Restlessness (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 7
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 12
Agitation (Psychiatric disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 6
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Lymphedema (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Hot Flashes (Vascular disorders) | 6
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT01540565/Prot_SAP_000.pdf